CLINICAL TRIAL: NCT00595972
Title: Phase II Trial of Epirubicin Cisplatin and FU Combined With Endostar in Patients With Advanced or Metastatic Gastric Cancer
Brief Title: Epirubicin Cisplatin and Fluorouracil (FU) Combined With Endostar in Patients With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Department of medical oncology, Cancer Hospital, Fuandan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECF/endo-MGC
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-09

CONDITIONS: Gastric Cancer
Keywords: Time to Progression; Overall survival; Response rate; Quality of Live; Toxicities
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): patients will be treated by ECF regimen (epirubicin, cisplatin plus 5-FU) combined with endostar
  Interventions: Drug: ECF-endostar

INTERVENTIONS:
Drug: ECF-endostar — Epirubicin 50mg/M2 D1, Cisplatin 60mg/M2 D1, FU 500mg/M2 D1-5, endostar 7.5mg/M2 D1-14, treatment cycle repeat every 3 weeks. Treatment should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Other Names: treatment group

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the ECF regimen (epirubicin, cisplatin and FU) combined with endostar-- a inhibitor of angiogenesis, in patients with advanced or metastatic gastric cancer (A/MGC).

DETAILED DESCRIPTION:
Although there is no standard regimen in the treatment of metastatic gastric cancer, ECF regimen (epirubicin, cisplatin and FU) is often considered as a reference regimen. And ECF regimen has been suggested as the first line therapy for A/MGC by FDA. According to the result of a Chinese phase III clinical trial in metastatic lung cancer, endostar-- a new angiogenesis inhibitor prolonged the overall survival, time to progression and improved response rate. So we designed this clinical trial to evaluate whether endostar can bring survival benefits to patients with advanced and metastatic gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* ECOG performance scale ≤ 2
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Adequate hepatic, renal, heart, and hematologic functions (platelets>80×109/L, neutrophil> 2.0 × 109/L, serum creatinine ≤ 1.5mg/dl, total bilirubin within upper limit of normal(ULN), and serum transaminase ≤ 2.5×the ULN)

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent cancer
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Neuropathy, brain, or leptomeningeal involvement
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or high risk/uncontrolled arrhythmia
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
time to progression | every two cycles

SECONDARY OUTCOMES:
toxicity | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China